CLINICAL TRIAL: NCT01882023
Title: Comparing Neural Responses to Explicit and Subliminal Food Images in EDNOS Patients and Healthy Controls Using fMRI
Brief Title: Comparing Neural Responses to Food Images in EDNOS Patients and Healthy Controls Using fMRI
Acronym: ANfMRI
Status: Recruiting | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: anfmri40
Record Dates: First submitted 2013-05-21; First posted 2013-06-20 (Estimated); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Eating Disorders
Keywords: EDNOS; adolescents; eating disorder; anorexia nervosa
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Eating disorder: Patients currently in treatment for eating disorders.
- Healthy Controls: Age- and gender matched healthy controls.

SUMMARY:
Currently, there is not a robust, testable neural model available that sufficiently explains the development and maintenance of anorexia nervosa (AN) a severe, often fatal, adolescent-onset eating disorder. Using state of the art neuroimaging and neuropsychological techniques, our objective is to identify neural mechanisms in the adolescent brain underlying AN. This is of high clinical relevance in as much as it will provide a robust platform for a diagnostic battery so that physicians can identify those who are prone to develop AN at a very early stage of life.

The aim of this research plan is: 1) To develop knowledge of cognitive dysfunction in adolescents who have recently been diagnosed with AN, with a battery of cognitive tests during a series of clinical visits. 2) To provide a scientific basis for our knowledge about how the brain of an adolescent with an eating disorder differs from that of a healthy adolescent, by conducting functional and structural magnetic resonance imaging on adolescent females with AN.

DETAILED DESCRIPTION:
Adolescents with eating disorders have debilitating cognitive disturbances that impact on their social, educational and physical health. One cognitive trait that is found to form core cognitive disturbances in AN is superior working memory (WM). WM is the ability to ruminate on a cognitive strategy while attending to the details of another task, excluding non-relevant stimuli, and is linked to activation of the dorsolateral prefrontal cortex (DLPFC). By administering functional Magnetic Resonance Imaging (fMRI) we have recently found that females with AN have increased activation in the DLPFC and reduced appetitive brain responses when thinking about eating food shown in visual images. This suggests that the increased WM capacity in AN may serve to suppress food intake, but this has not yet been clarified. In line with this assumption, we have also shown that restraint of appetite in those with AN was linked to greater plasticity in the DLPFC. Furthermore, Transcranial Magnetic Stimulation (TMS) of the DLPFC reduces appetitive responses to food stimuli in adults with eating disorders. Conversely, we have shown that being obese is linked to reduced structure and abnormal function in the DLPFC, as well as reduced attentional control/WM performance. Therefore, it is likely that DLPFC-related WM function is associated with eating disorders, particularly cognitive restraint of appetite.

It is likely that the interaction between appetitive brain regions and specific prefrontal cortex (PFC) cognitions determines whether an adolescent develops anorexia nervosa. We aim to provide neuropsychological and brain imaging measures showing how a specific cognitive function is linked to early-onset disordered eating behaviour, and we will do this before and after standard clinical treatment. We suggest that such understanding could enable school nurses to use the unique paradigm we use in our fMRI study, to detect illness before it damages the child's life and becomes difficult to treat.

The study has now been increased to include genetic components to examine the genetic and epigenetic variation for genes found to be linked with eating disorders.

ELIGIBILITY:
Inclusion Criteria:

* Females
* Age 13 - 18 yrs
* Right handed
* For controls: BMI within the "normal" range
* For patients: Be admitted to treatment for an eating disorder

Exclusion Criteria:

* On medication
* Suffering from any other illnesses
* Left handed
* Metal implants which can impact the fMRI image
* Severe claustrophobia
* Pregnancy
* Smoker
* Regular alcohol drinker

Ages: 13 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Half of the cohort are patients recruited from the eating disorder clinic. All subjects in the study are adolescent females residing in the Uppsala area.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2011-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Measure functional differences in adolescents with eating disorders and healthy controls. | This is measured during scanning shortly after patient admittance to treatment, and one year later. Controls have their scans shortly after being recruited to the study, then again 1 year later.
  The analysis of each groups' neural activity will be carried out with statistical parametric mapping (SPM) implemented in Matlab. This will compare the statistical parametric maps between the group using ANOVAs, ANCOVAs and t-tests.

SECONDARY OUTCOMES:
Measure structural differences in adolescents with eating disorders and healthy controls. | This is measured during scanning shortly after patient admittance to treatment, and one year later. Controls have their scans shortly after being recruited to the study, then again 1 year later.
  To determine any structural differences, matlab will be used. With this one can upload the T1 structural scanning data and determine the volume of each subject's brain, and even compute the volume of each tissue (CBF, white matter and grey matter).
Develop knowledge of cognitive dysfunction in adolescents with eating disorders. | The cognitive measures are conducted shortly after recruitment of the study. The subjects are given the questionnaires upon their first meeting, and are posted back to us shortly after.
  Any cognitive dysfunction will be measured with a working memory task in the scanner (N-back task). Further, various clinical variables will be measured with the use of questionnaires such as Eating Disorder Examination Questionnaire (EDEQ), Perceived Stress Scale (PSS), Montgomery-Åsberg Depression Rate Scale (MADRS), Eating Disorder Inventory (EDI), Barratts Impulsivity Scale (BIS), Obsessive Compulsive Inventory - Revised (OCI R), and Multidimensional Perfectionism Scale (MPS).
To examine whether clinical variables can predict neural activity. | The neural activity is measured during scanning shortly after subject recruitment, and one year later. The clinical measurements are measured with questionnaires given to them on their first meeting after recruitment, which are later posted back to us.
  The analysis of each groups' neural activity will be carried out with statistical parametric mapping (SPM) implemented in Matlab. This will compare the statistical parametric maps between the group using ANOVAs, ANCOVAs and t-tests. The clinical variables will be measured with the use of questionnaires such as Eating Disorder Examination Questionnaire (EDEQ), Perceived Stress Scale (PSS), Montgomery-Åsberg Depression Rate Scale (MADRS), Eating Disorder Inventory (EDI), Barratts Impulsivity Scale (BIS), Obsessive Compulsive Inventory - Revised (OCI R), and Multidimensional Perfectionism Scale (MPS). These will be used in a multiple regression analysis carried out in SPM to see whether there is any correlation between the scores of the questionnaires and the brain activity of the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Zhukovsky, MMed, Principal Investigator — Uppsala University
Locations (1):
- Röntgenavdelningen, Uppsala Academic Hospital, Uppsala, Uppsala County, Sweden

REFERENCES:
- [Background] Brooks SJ, O'Daly OG, Uher R, Schioth HB, Treasure J, Campbell IC. Subliminal food images compromise superior working memory performance in women with restricting anorexia nervosa. Conscious Cogn. 2012 Jun;21(2):751-63. doi: 10.1016/j.concog.2012.02.006. Epub 2012 Mar 11. PMID 22414738
- [Background] Andrews SC, Hoy KE, Enticott PG, Daskalakis ZJ, Fitzgerald PB. Improving working memory: the effect of combining cognitive activity and anodal transcranial direct current stimulation to the left dorsolateral prefrontal cortex. Brain Stimul. 2011 Apr;4(2):84-9. doi: 10.1016/j.brs.2010.06.004. Epub 2010 Jul 11. PMID 21511208
- [Background] Brooks SJ, O'Daly OG, Uher R, Friederich HC, Giampietro V, Brammer M, Williams SC, Schioth HB, Treasure J, Campbell IC. Differential neural responses to food images in women with bulimia versus anorexia nervosa. PLoS One. 2011;6(7):e22259. doi: 10.1371/journal.pone.0022259. Epub 2011 Jul 20. PMID 21799807
- [Background] Brooks SJ, O'Daly O, Uher R, Friederich HC, Giampietro V, Brammer M, Williams SC, Schioth HB, Treasure J, Campbell IC. Thinking about eating food activates visual cortex with reduced bilateral cerebellar activation in females with anorexia nervosa: an fMRI study. PLoS One. 2012;7(3):e34000. doi: 10.1371/journal.pone.0034000. Epub 2012 Mar 27. PMID 22479499
- [Background] Brooks SJ, Barker GJ, O'Daly OG, Brammer M, Williams SC, Benedict C, Schioth HB, Treasure J, Campbell IC. Restraint of appetite and reduced regional brain volumes in anorexia nervosa: a voxel-based morphometric study. BMC Psychiatry. 2011 Nov 17;11:179. doi: 10.1186/1471-244X-11-179. PMID 22093442
- [Background] Van den Eynde F, Claudino AM, Mogg A, Horrell L, Stahl D, Ribeiro W, Uher R, Campbell I, Schmidt U. Repetitive transcranial magnetic stimulation reduces cue-induced food craving in bulimic disorders. Biol Psychiatry. 2010 Apr 15;67(8):793-5. doi: 10.1016/j.biopsych.2009.11.023. Epub 2010 Jan 8. PMID 20060105
- [Background] Brooks SJ, Benedict C, Burgos J, Kempton MJ, Kullberg J, Nordenskjold R, Kilander L, Nylander R, Larsson EM, Johansson L, Ahlstrom H, Lind L, Schioth HB. Late-life obesity is associated with smaller global and regional gray matter volumes: a voxel-based morphometric study. Int J Obes (Lond). 2013 Feb;37(2):230-6. doi: 10.1038/ijo.2012.13. Epub 2012 Jan 31. PMID 22290540
- [Background] Olivo G, Wiemerslage L, Swenne I, Zhukovsky C, Salonen-Ros H, Larsson EM, Gaudio S, Brooks SJ, Schioth HB. Correction: Limbic-thalamo-cortical projections and reward-related circuitry integrity affects eating behavior: A longitudinal DTI study in adolescents with restrictive eating disorders. PLoS One. 2017 Apr 20;12(4):e0176646. doi: 10.1371/journal.pone.0176646. eCollection 2017. PMID 28426755
- [Background] Olivo G, Wiemerslage L, Swenne I, Zhukowsky C, Salonen-Ros H, Larsson EM, Gaudio S, Brooks SJ, Schioth HB. Limbic-thalamo-cortical projections and reward-related circuitry integrity affects eating behavior: A longitudinal DTI study in adolescents with restrictive eating disorders. PLoS One. 2017 Mar 1;12(3):e0172129. doi: 10.1371/journal.pone.0172129. eCollection 2017. PMID 28248991
- [Background] Olivo G, Zhou W, Sundbom M, Zhukovsky C, Hogenkamp P, Nikontovic L, Stark J, Wiemerslage L, Larsson EM, Benedict C, Schioth HB. Resting-state brain connectivity changes in obese women after Roux-en-Y gastric bypass surgery: A longitudinal study. Sci Rep. 2017 Jul 26;7(1):6616. doi: 10.1038/s41598-017-06663-5. PMID 28747648
- [Background] Gaudio S, Carducci F, Piervincenzi C, Olivo G, Schioth HB. Altered thalamo-cortical and occipital-parietal- temporal-frontal white matter connections in patients with anorexia and bulimia nervosa: a systematic review of diffusion tensor imaging studies. J Psychiatry Neurosci. 2019 Sep 1;44(5):324-339. doi: 10.1503/jpn.180121. PMID 30994310
- [Background] Olivo G, Swenne I, Zhukovsky C, Tuunainen AK, Saaid A, Salonen-Ros H, Larsson EM, Brooks SJ, Schioth HB. Preserved white matter microstructure in adolescent patients with atypical anorexia nervosa. Int J Eat Disord. 2019 Feb;52(2):166-174. doi: 10.1002/eat.23012. Epub 2019 Jan 24. PMID 30676658
- [Background] Olivo G, Swenne I, Zhukovsky C, Tuunainen AK, Salonen-Ros H, Larsson EM, Gaudio S, Brooks SJ, Schioth HB. Reduced resting-state connectivity in areas involved in processing of face-related social cues in female adolescents with atypical anorexia nervosa. Transl Psychiatry. 2018 Dec 13;8(1):275. doi: 10.1038/s41398-018-0333-1. PMID 30546060
- [Background] Gaudio S, Olivo G, Beomonte Zobel B, Schioth HB. Altered cerebellar-insular-parietal-cingular subnetwork in adolescents in the earliest stages of anorexia nervosa: a network-based statistic analysis. Transl Psychiatry. 2018 Jul 6;8(1):127. doi: 10.1038/s41398-018-0173-z. PMID 29980676
- [Background] Olivo G, Solstrand Dahlberg L, Wiemerslage L, Swenne I, Zhukovsky C, Salonen-Ros H, Larsson EM, Gaudio S, Brooks SJ, Schioth HB. Atypical anorexia nervosa is not related to brain structural changes in newly diagnosed adolescent patients. Int J Eat Disord. 2018 Jan;51(1):39-45. doi: 10.1002/eat.22805. Epub 2017 Dec 7. PMID 29215777